CLINICAL TRIAL: NCT02121054
Title: Research of Resistance to Antiplatelet Agents and Development of Tailored Treatment Model for Patients With Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: Young-Hak Kim, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Young-Hak Kim, MD, PhD, MD, PhD, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: 2013-0873
Record Dates: First submitted 2014-04-21; First posted 2014-04-23 (Estimated); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Cardiovascular Diseases; Coronary Artery Disease
Keywords: Antiplatelet Agents; Drug Resistance
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the prognosis of patients with resistance to antiplatelet agent and develop tailored treatment model for patients with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Age >20
* Patients with coronary artery disease
* Patients with peripheral artery disease

Exclusion Criteria:

* Renal dysfunction
* Hepatic dysfunction
* Major surgery planned within 1 year
* Malignant tumor
* History of gastrointestinal bleeding
* low or high platelet count

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease, Patients with peripheral artery disease
Sampling Method: Probability Sample
Enrollment: 1527 (Actual)
Dates: Start 2013-10-19 (Actual); Primary Completion 2020-10-29 (Actual); Study Completion 2020-10-29 (Actual)

PRIMARY OUTCOMES:
Major adverse event | 2 year
  Major adverse event : overall mortality, cardiovascular mortality, target vessel revascularization

SECONDARY OUTCOMES:
Biomarker | 2 year
  homocysteine, Lp(a), fibrinogen, PAI-1, NTpro-BNP, hs-CRP, matrix metalloproteinase-9, soluble CD40L, IL-6, serum amyloid A, AGE

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Songpa-Gu, South Korea